CLINICAL TRIAL: NCT03489590
Title: 19F Magnetic Resonance Imaging to Evaluate Regional Ventilation in Healthy Subjects and Subjects With Cystic Fibrosis
Brief Title: 19F MRI to Evaluate Regional Ventilation in Healthy Subjects and Subjects With Cystic Fibrosis
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 14-0509
Record Dates: First submitted 2018-03-29; First posted 2018-04-05 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: Cystic Fibrosis
Keywords: Lung; Imaging; Hyperpolarized; Perfluorinated; MRI
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Intervention Model Description: This study enrolls both healthy volunteers and volunteers with cystic fibrosis. Both healthy and CF participants will receive the same treatment throughout the entirety of the study.
Oversight: Data Monitoring Committee: No

ARMS (1):
- 19F MRI with PFP (Experimental): PFP gas will be administered using a full-face mask during the MRI. Images are acquired during 12-second breath-hold after every 3rd breath. Before and after the MRI is complete, participants will perform spirometry maneuvers in a room outside of the magnet.
  Interventions: Drug: PFP

INTERVENTIONS:
Drug: PFP — * Composition: inhaled PFP, a gaseous contrast agent (79% PFP, 21% O2, pre-mixed, medical grade gas)
  * Administration: Full-face disposable ventilation mask and a standard Douglas Bag system.
  * Dosage: Two controlled breaths of contrast gas followed by a full breath and a 12-second breath-hold and scan for image acquisition.
  * Frequency: Repeated 5 times followed by an identical five cycles with room air to ensure PFP gas wash-out has occurred.
  Other Names: Perfluoropropane gas (C3F8); 19F

SUMMARY:
An open label non-randomized study enrolling up to 20 healthy participants and up to 30 participants with cystic fibrosis to establish a healthy versus disease comparison. Each participant will receive a mixture of inert gas (perfluoropropane (PFP)) in a ratio of 79% PFP to 21% oxygen as a contrast agent to enhance visualization of the airway and alveolar spaces using magnetic resonance imaging of inert gas/oxygen mixtures. The study consists of a screening visit followed by up to 2 study visits.

DETAILED DESCRIPTION:
The goal of this study is to evaluate the ability of conventional 'thermally' polarized perfluorinated gases (19F) mixed with oxygen to detect changes in ventilation using magnetic resonance imaging (MRI). A secondary goal is to assess the repeatability and the within-subject variability of these findings in CF lung disease. This is an open label pilot study expanding on work by other investigators currently using this technique in human subjects. Projection images using controlled breathing techniques will be obtained using 19F MRI, correlating spirometric variables with regional distribution of the gases.

ELIGIBILITY:
Inclusion Criteria for Healthy Participants:

* Non-smokers (<10 pack-year history, and no active smoking in last 1 year);
* No evidence of prior lung disease or lung injury by medical history, physical exam, and/or spirometry testing;
* Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the trial.
* Participants must be willing and able to comply with scheduled visits and other trial procedures.

Exclusion Criteria for Healthy Participants:

* Active or past smokers with less than 1 years since quitting or >10 pack-year smoking history
* Unable to undergo a 3.0-Tesla MRI exam of the lungs and chest because of contraindications including

  1. Occupation (past or present) of machiner, welder, grinder;
  2. Injury to the eye involving a metallic object
  3. Injury to the body by a metallic object (bullet, BB, shrapnel)
  4. Presence of a cardiac pacemaker or defibrillator
  5. Presence of aneurysm clips
  6. Presence of carotid artery vascular clamp
  7. Presence of neurostimulator
  8. Presence of insulin or infusion pump
  9. Presence of implanted drug infusion device that is not known to be MRI compatible (i.e., was placed outside of UNCH or is older than 10 years)
  10. Bone growth or fusion simulator
  11. Presence of cochlear, otologic or ear implant
  12. Any type of prosthesis (eye, penile, etc.)
  13. Artificial limb or joint
  14. Non-removable electrodes (on body, head or brain)
  15. Intravascular stents, filters or coils
  16. Shunt (spinal or intraventricular)
  17. Swan-ganz catheter
  18. Any implant held in place by a magnet
  19. Transdermal delivery system (e.g. Nitro)
  20. IUD or diaphragm
  21. Tattooed makeup (eyeliner, lips, etc.) or tattoos covering >25% of body surface area
  22. Body piercings (MUST BE REMOVED BEFORE MRI)
  23. Any metal fragments
  24. Internal pacing wires
  25. Metal or wire mesh implants
  26. Hearing aid (REMOVE BEFORE MRI) aa. Dentures (REMOVE BEFORE MRI) bb. Claustrophobia
* Unable to tolerate inhalation of gas mixture
* Participation in a clinical trial with a study drug that may impact lung function in the past 14 days
* Other severe acute or chronic medical or psychiatric condition or clinical laboratory abnormality that may increase the risk associated with trial participation or may interfere with the interpretation of trial results and, in the judgment of the investigator, would make the participant inappropriate for entry into this trial.
* Pregnancy: women of childbearing potential must have a confirmed negative urine pregnancy test on the day of the MR scan, prior to the MRI scan.

Inclusion Criteria for CF Participants:

* Non-smokers (<10 pack year history and no active smoking in the past year;
* Diagnosis of cystic fibrosis as via standard sweat chloride/phenotypic features/genotyping
* Stable lung disease as evidenced by no change in respiratory medications or change in FEV1 of >15% from baseline over the preceding 4 weeks prior to enrollment
* Baseline FEV1 >30% of predicted. Roughly equivalent numbers of CF subjects with mild FEV1 >80% of predicted), moderate (FEV1 50-80% of predicted) and severe (FEV1 <50% of predicted) will be targeted for enrollment.
* No use of supplemental oxygen
* Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the trial.
* Participants must be willing and able to comply with scheduled visits and other trial procedures.

Exclusion Criteria for CF Participants:

* Active or past smokers with less than 1 years since quitting or >10 pack-year smoking history
* Active asthma flare, as perceived by the study physician or unstable asthma characterized by advancement of asthma therapy in the last month or two courses of oral steroids in the past six months.
* Unable to undergo a 3.0-Tesla MRI exam of the lungs and chest because of contraindications including

  1. Occupation (past or present) of machiner, welder, grinder;
  2. Injury to the eye involving a metallic object
  3. Injury to the body by a metallic object (bullet, BB, shrapnel)
  4. Presence of a cardiac pacemaker or defibrillator
  5. Presence of aneurysm clips
  6. Presence of carotid artery vascular clamp
  7. Presence of neurostimulator
  8. Presence of insulin or infusion pump
  9. Presence of implanted drug infusion device that is not known to be MRI compatible (i.e., was placed outside of UNCH or is older than 10 years)
  10. Bone growth or fusion simulator
  11. Presence of cochlear, otologic or ear implant
  12. Any type of prosthesis (eye, penile, etc.)
  13. Artificial limb or joint
  14. Non-removable electrodes (on body, head or brain)
  15. Intravascular stents, filters or coils
  16. Shunt (spinal or intraventricular)
  17. Swan-ganz catheter
  18. Any implant held in place by a magnet
  19. Transdermal delivery system (e.g. Nitro)
  20. IUD or diaphragm
  21. Tattooed makeup (eyeliner, lips, etc.) or tattoos covering >25% of body surface area
  22. Body piercings (MUST BE REMOVED BEFORE MRI)
  23. Any metal fragments
  24. Internal pacing wires
  25. Metal or wire mesh implants
  26. Hearing aid (REMOVE BEFORE MRI) aa. Dentures (REMOVE BEFORE MRI) bb. Claustrophobia
* Unable to tolerate inhalation of gas mixture
* Participation in a clinical trial with a study drug that may impact lung function in the past 14 days
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with trial participation or may interfere with the interpretation of trial results and, in the judgment of the investigator, would make the participant inappropriate for entry into this trial.
* Pregnancy; women of childbearing potential must have a confirmed negative urine pregnancy test on the day of the MR scan, prior to the MRI scan.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Obtain technically sufficient 19F MRI images | 1 day
  Determine if 19F gas images of the human lung and airways can be obtained in both single breath-hold and gated breathing imaging studies with adequate signal level and image contrast to extract regional lung ventilation information.

SECONDARY OUTCOMES:
Determine the reproducibility of ventilation assessments in the adult cystic fibrosis (CF) population. | 1 week
  Repeated scans will be optional for CF participants in order to begin to understand the repeatability of this outcome measure
Compare quantitative and qualitative image measures of lung ventilation using 19F MRI imaging to spirometric values. | 1 day
  Pair 19F lung images and Ventilation Defect Percentages with FEV1 obtained via spirometry

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L Goralski, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Couch MJ, Ball IK, Li T, Fox MS, Littlefield SL, Biman B, Albert MS. Pulmonary ultrashort echo time 19F MR imaging with inhaled fluorinated gas mixtures in healthy volunteers: feasibility. Radiology. 2013 Dec;269(3):903-9. doi: 10.1148/radiol.13130609. Epub 2013 Oct 28. PMID 23985278
- [Background] Halaweish AF, Moon RE, Foster WM, Soher BJ, McAdams HP, MacFall JR, Ainslie MD, MacIntyre NR, Charles HC. Perfluoropropane gas as a magnetic resonance lung imaging contrast agent in humans. Chest. 2013 Oct;144(4):1300-1310. doi: 10.1378/chest.12-2597. PMID 23722696
- [Derived] Goralski JL, Chung SH, Glass TM, Ceppe AS, Akinnagbe-Zusterzeel EO, Trimble AT, Boucher RC, Soher BJ, Charles HC, Donaldson SH, Lee YZ. Dynamic perfluorinated gas MRI reveals abnormal ventilation despite normal FEV1 in cystic fibrosis. JCI Insight. 2020 Jan 30;5(2):e133400. doi: 10.1172/jci.insight.133400. PMID 31855577